CLINICAL TRIAL: NCT01865175
Title: A Pilot Study Comparing Tolerance of Oral Heme Iron Polypeptide With Oral Ionic Iron
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Institution required IND, although FDA did not, so institution did not allow enrollment
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Andrew S. Freiberg, Associate Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HIP ASF1
Record Dates: First submitted 2013-05-26; First posted 2013-05-30 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ionic iron (Active Comparator): Subjects will take ionic iron daily for 7 days followed by 7 days of no medicine folloowed by 7 days of heme iron.
  Interventions: Drug: ionic iron; Drug: heme iron polypeptide
- heme iron polypeptide (Experimental): Subject will take heme iron daily for 7 days followed by 7 days of no medicine followed by 7 days of ionic iron.
  Interventions: Drug: ionic iron; Drug: heme iron polypeptide

INTERVENTIONS:
Drug: ionic iron — Subjects will take ionic iron daily for 7 days followed by 7 days of no medicine followed by 7 days of heme iron.
  Other Names: Ferrous Sulphate
Drug: heme iron polypeptide — Subject will take heme iron daily for 7 days followed by 7 days of no medicine followed by 7 days of ionic iron.
  Other Names: Proferrin; HIP

SUMMARY:
This is a pilot study designed to compare the tolerance of ionic iron (ferrous sulphate) with heme iron polypeptide. Subjects will take one week of one product followed by a week with no product followed by a week with the other product. Subjects will complete a daily diary to assess side effects.

Hypothesis: Heme iron polypeptide is associated with fewer gastrointestinal side effects than ionic iron.

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) is a worldwide problem in both children and adults. Traditional ionic oral iron supplements have many disadvantages including high gastrointestinal side effects, poor and variable absorption, poor compliance, and the potential for overdose, especially in children. Proferrin is a currently available form of heme iron polypeptide (HIP). It is different from older more traditional iron formulations, such as ferrous sulphate, in that it is heme iron as opposed to ionic iron. The porphyrin ring of heme allows the iron to be absorbed through a different receptor than ionic iron resulting in different absorption kinetics and GI side effect profiles. The absorption of HIP is via the same mechanism as dietary iron contained in meat. Therefore, heme iron therapy may avoid several problems associated with ionic iron therapy such as gastrointestinal side effects and absorption that is dependent on food intake.

30 subjects will be enrolled, randomized to starting with one or the other study drug, but crossing over to the other, so that all subjects will be in a single cohort. This is an open label randomized pilot study intended to test the feasibility of collecting information on drug tolerance. The randomization will be stratified by age, gender and hemoglobin.

An optional baseline blood test will be drawn (CBC, iron profile, ferritin). If subjects decide to participate in the optional blood draws, they will return during the week they are not taking either study medication for this test. For subjects not participating in the optional blood tests and not needing to return to the clinic for another reason, subjects will be contacted by phone (or in person if returning to the clinic for another reason) during the week not taking either medication to address any concerns or issues. If not agreeing to participate in the blood tests, they will be allowed to send the empty pill bottles and the diary by mail and will be contacted by phone to make sure there were no problems during the study. If participating in the optional blood tests, within one month after taking the final pill, subjects will return to the clinic to return the medication containers and study diary.

ELIGIBILITY:
Inclusion Criteria:

* able to fill out daily diary

Exclusion Criteria:

* known iron overload
* sensitivity to either product used

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
tolerance | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Freiberg, M.D., Principal Investigator — Penn State University
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States